CLINICAL TRIAL: NCT01106820
Title: Progressive Resistance Training vs. Relaxation for Breast Cancer Patients During Chemotherapy: A Randomized Controlled Intervention Trial to Evaluate the Biological Mechanisms and Effects of Resistance Training on Fatigue and Quality of Life
Brief Title: Progressive Resistance Training Versus Relaxation for Breast Cancer Patients During Chemotherapy: Biological Mechanisms and Effects on Fatigue and Quality of Life
Acronym: BEATE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: German Cancer Research Center (Other)
Collaborators: National Center for Tumor Diseases, Heidelberg (Other); University Hospital Heidelberg (Other); Central Institute of Mental Health, Mannheim (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BEATE-1
Record Dates: First submitted 2010-04-14; First posted 2010-04-20 (Estimated); Last update posted 2016-12-19 (Estimated); Status verified 2016-12

CONDITIONS: Breast Cancer; Cancer-related Fatigue
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Resistance training (Active Comparator)
  Interventions: Other: Supervised progressive resistance training
- Relaxation training (Active Comparator)
  Interventions: Other: Supervised progressive muscle relaxation training (Jacobsen method)

INTERVENTIONS:
Other: Supervised progressive resistance training — Supervised progressive resistance training
  Arms: Resistance training
Other: Supervised progressive muscle relaxation training (Jacobsen method) — Supervised progressive muscle relaxation training (Jacobsen method)
  Arms: Relaxation training

SUMMARY:
The purpose of this randomized intervention study is to investigate the effects and biological mechanisms of a supervised 12-week progressive resistance training on fatigue and quality of life in breast cancer patients during chemotherapy. To determine the effect of the exercise itself beyond potential psychosocial effects due to attention by trainers or the group support, patients in the control group have a comparable training schedule (i.e. 60 min, twice a week, for 12 weeks) but with relaxation training (Jacobsen method).

ELIGIBILITY:
Inclusion Criteria:

* breast cancer patient after lumpectomy or mastectomy, stage I-III
* adjuvant chemotherapy
* BMI at least 18

Exclusion Criteria:

* contraindication for exercise
* radiotherapy during intervention period

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2010-04; Primary Completion 2013-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Fatigue measured by Fatigue Assessment Questionnaire (FAQ) | change between baseline and week 13 (end of intervention)

SECONDARY OUTCOMES:
Quality of Life measured by the European Organisation for Research and Treatment of Cancer questionnaire (EORTC-QLQ30/BR23) | change between baseline and week 13 (end of intervention)
Depression measured by "Allgemeine Depressionsskala" (ADS, the German version of the Center for Epidemiological Studies Depression Scale (CES-D)) | change between baseline and week 13 (end of intervention)
Muscle strength measured at the IsoMed2000® | change between baseline and week 13 (end of intervention)
Cardiorespiratory fitness measured by ergospirometry | change between baseline and week 13 (end of intervention)
Biomarker in blood, urine, and saliva | change between baseline and week 6 and 13
Number of patients with adverse events potentially related to the resistance training | during the 12-week exercise intervention

CONTACTS AND LOCATIONS:
Overall Officials: Karen Steindorf, Prof. Dr., Principal Investigator — NCT Heidelberg
Locations (1):
- German Cancer Research Center, Heidelberg, Germany

REFERENCES:
- [Background] Schmidt ME, Wiskemann J, Krakowski-Roosen H, Knicker AJ, Habermann N, Schneeweiss A, Ulrich CM, Steindorf K. Progressive resistance versus relaxation training for breast cancer patients during adjuvant chemotherapy: design and rationale of a randomized controlled trial (BEATE study). Contemp Clin Trials. 2013 Jan;34(1):117-25. doi: 10.1016/j.cct.2012.10.006. Epub 2012 Oct 25. PMID 23103936
- [Result] Schmidt ME, Wiskemann J, Armbrust P, Schneeweiss A, Ulrich CM, Steindorf K. Effects of resistance exercise on fatigue and quality of life in breast cancer patients undergoing adjuvant chemotherapy: A randomized controlled trial. Int J Cancer. 2015 Jul 15;137(2):471-80. doi: 10.1002/ijc.29383. Epub 2014 Dec 16. PMID 25484317
- [Result] Klassen O, Schmidt ME, Scharhag-Rosenberger F, Sorkin M, Ulrich CM, Schneeweiss A, Potthoff K, Steindorf K, Wiskemann J. Cardiorespiratory fitness in breast cancer patients undergoing adjuvant therapy. Acta Oncol. 2014 Oct;53(10):1356-65. doi: 10.3109/0284186X.2014.899435. Epub 2014 May 16. PMID 24837860
- [Result] Scharhag-Rosenberger F, Kuehl R, Klassen O, Schommer K, Schmidt ME, Ulrich CM, Wiskemann J, Steindorf K. Exercise training intensity prescription in breast cancer survivors: validity of current practice and specific recommendations. J Cancer Surviv. 2015 Dec;9(4):612-9. doi: 10.1007/s11764-015-0437-z. Epub 2015 Feb 26. PMID 25711667
- [Derived] Koeppel M, Steindorf K, Schmidt ME, Rosenberger F, Wiskemann J. Variability in resistance training trajectories of breast cancer patients undergoing therapy. Support Care Cancer. 2024 Dec 10;33(1):12. doi: 10.1007/s00520-024-09001-4. PMID 39656317
- [Derived] Ernst M, Wagner C, Oeser A, Messer S, Wender A, Cryns N, Brockelmann PJ, Holtkamp U, Baumann FT, Wiskemann J, Monsef I, Scherer RW, Mishra SI, Skoetz N. Resistance training for fatigue in people with cancer. Cochrane Database Syst Rev. 2024 Nov 28;11(11):CD015518. doi: 10.1002/14651858.CD015518. PMID 39606939
- [Derived] Schmidt ME, Wiskemann J, Johnson T, Habermann N, Schneeweiss A, Steindorf K. L-Thyroxine intake as a potential risk factor for the development of fatigue in breast cancer patients undergoing chemotherapy. Support Care Cancer. 2018 Aug;26(8):2561-2569. doi: 10.1007/s00520-018-4095-3. Epub 2018 Feb 14. PMID 29445858